CLINICAL TRIAL: NCT02840552
Title: The Safety and Efficacy of 18F-Fluoromethylcholine (18F-FCH) PET/CT in Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Stephan Probst, Chief of Nuclear Medicine, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-061
Record Dates: First submitted 2016-07-14; First posted 2016-07-21 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluoromethylcholine; fluorocholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FCH-PET/CT (Experimental): 18F-Fluoromethylcholine (18F-FCH) PET/CT
  Interventions: Drug: 18F-Fluoromethylcholine (18F-FCH)

INTERVENTIONS:
Drug: 18F-Fluoromethylcholine (18F-FCH) — FCH PET/CT

SUMMARY:
The objectives of this study are to confirm the safety and efficacy of FCH-PET/CT and to establish our ability to reproduce results from the literature using FCH-PET/CT as a diagnostic and decision making tool in the management in two predefined groups of prostate cancer patients, specifically, biochemical recurrence and high risk staging. The primary endpoints of the study are the incidence of adverse events (AE) in the study population up to 24 hours following the scan, and the sensitivity and specificity of FCH-PET/CT vs CT on a per-patient and per-lesion basis.

DETAILED DESCRIPTION:
Background Prostate cancer is the second leading cause of cancer death in North American men older than 50 years. Positron emission tomography / computer tomography (PET/CT) is a nuclear medicine procedure based on the measurement of positron emission from radiolabeled tracer molecules. A common radiotracer in use today is 18F-fluoromethylcholine (aka fluorocholine or FCH) which is a radiolabeled choline derivative. Imaging with FCH-PET/CT can be used to characterize and localize prostate cancer in vivo. There is extensive data in the literature showing the value of FCH-PET/CT imaging in accurately staging and restaging prostate cancer. FCH-PET/CT is standard of care in many European countries.

Study Objectives The objectives of this study are to confirm the safety and efficacy of FCH-PET/CT and to establish our ability to reproduce results from the literature using FCH-PET/CT as a diagnostic and decision making tool in the management in two predefined groups of prostate cancer patients, specifically, biochemical recurrence and high risk staging. The primary endpoints of the study are the incidence of adverse events (AE) in the study population up to 24 hours following the scan, and the sensitivity and specificity of FCH-PET/CT vs CT on a per-patient and per-lesion basis.

Study Design This will be a multi-center open label study in which one (1) FCH-PET/CT will be performed on study participants. A PET/CT scan takes 2-3 hours.

Safety FCH-PET/CT exhibits favorable dosimetry, delivering organ doses that are comparable to or lower than those delivered by 18F-FDG. The safety of FCH is not disputed and we expect the number of adverse events in our study to be zero.

Sample Size and Recruitment Target enrollment is 1500 patients. This will be sufficient to detect AE with a prevalence of 0.3% with 99% confidence. For efficacy endpoints, approximately 500 subjects would provide 90% power at the alpha=0.05 one-sided level of significance that the specificity and sensitivity will be superior to the specificity and sensitivity under the null hypothesis. Patients will be recruited by urologists in the clinical setting. Initial contact and consent will be by the department of urology.

ELIGIBILITY:
Global Inclusion Criteria:

* Resident of Canada
* Male sex
* Age 18 years or older
* Previously diagnosed with prostate cancer, under referring physician's care
* ECOG performance status 0 - 3, inclusive
* Able to understand and provide written informed consent
* Able to tolerate the physical/logistical requirements of completing a PET/CT scan including lying supine (or prone) for up to 40 minutes and tolerating intravenous cannulation for injection

Global Exclusion Criteria:

* Patients who are medically unstable (e.g. acute cardiac or respiratory distress or hypotensive)
* Patients who exceed the safe weight limit of the PET/CT bed (usually approximately 400 lbs.) or who cannot fit through the PET/CT bore (usually approximately 70 cm diameter)
* Patients who are claustrophobic.

Clinical Indication Criteria Subgroups:

* BCR: Biochemical recurrence as defined by serum PSA > 1 ng/ml following either radical prostatectomy or curative-intent radiotherapy or other prostate-ablative definitive management.
* HRS: Staging of high risk patients as defined by any one of the following:

  * Gleason score > 7
  * Serum PSA > 15 ng/ml
  * T stage of T3 or greater on TNM staging
  * Equivocal conventional staging such as CT, MRI or bone scan
  * Clinical suspicion of advance stage disease (e.g. bone pain)

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety of FCH-PET/CT imaging as measured by the incidence of adverse events (AE) | 7 days
Efficacy of FCH-PET/CT imaging as measured by sensitivity and specificity vs CT on a per patient basis as compared to standard of truth | 12 months
Efficacy of FCH-PET/CT imaging as measured by sensitivity and specificity vs CT on a per lesion basis as compared to standard of truth | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada